CLINICAL TRIAL: NCT00945126
Title: Allogeneic Stem Cell Transplantation With CD3/CD19 Depleted Stem Cells of Related or Unrelated Haploidentical Donors in Pediatric Patients With Malignant and Non-malignant Diseases
Brief Title: Allogeneic Stem Cell Transplantation in Pediatric Patients With Malignant and Non-malignant High-risk Diseases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrural
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Peter Bader, Prof. Dr. med. Peter Bader, Johann Wolfgang Goethe University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZKI-SCT-HAPLO-0106
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Malignant and Non-malignant High Risk Diseases
Keywords: Allogeneic stem cell transplantation in pediatric patients; CD3/CD19 depleted stem cells; malignant and non-malignant high risk diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Hematopoietic stem cell product from haploidentical or unrelated donor CD3/CD19 depleted with CliniMACS — The aim is to transplant 7x106 CD34+/kg of recipient body weight.

SUMMARY:
The aim of the study is to investigate the feasibility and toxicity of allogeneic haploidentical or unrelated transplantation with CD3/CD19 depleted stem cells associated with a reduced or a standard conditioning regimen in pediatric patients with malignant and non-malignant high-risk diseases, for whom allogeneic stem cell transplantation represents the only possible therapy option and no human leukocyte antigen (HLA) compatible related donors are available.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 0 to 30 years
* Written informed consent from patient and/or parents or guardian
* Patients with Karnofsky Index > 60%
* Malignant disease:

  * acute lymphoblastic leukemia
  * acute myeloid leukemia
  * myelodysplastic syndrome
  * chronic myeloid leukemia according to the standard indications
  * solid tumors (e.g. neuroblastoma recurrence, soft-tissue sarcoma, Ewing's sarcoma, osteosarcoma, hepatoblastoma)

    . Non malignant disease:
  * acquired anemias (e.g. severe aplastic anemia, particularly severe Evans syndrome)
  * congenital anemias (e.g. thalassemia and sickle cell anemia)
* Women reliable contraception method when appropriate

Exclusion Criteria:

* Participation in other clinical trials
* Patients, parents, or guardians unable to understand the nature, the importance and the implications of the procedure
* Pregnant or nursing women
* Patients who underwent a stem cell transplantation in the last 250 days
* Patients with kidney, heart or liver insufficiency

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2006-12; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
To evaluate engraftment after CD3/CD19 depletion of the graft | within 1 year

SECONDARY OUTCOMES:
To evaluate immunoreconstitution after transplantation by assessing lymphocyte subsets | within 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bader, Professor, Principal Investigator — University Hospital Frankfurt, Dept. for Children and Adolescents, Division for Stem Cell Transplantation, Goethe University.
Locations (1):
- University Hospital Frankfurt, Dept. for Children and Adolescents, Division for Stem Cell Transplantation, Goethe University, Frankfurt am Main, Hesse, Germany